CLINICAL TRIAL: NCT04070261
Title: Usability Comparison of a mHealth Application for Pre-anesthesia Evaluation Before and After Re-design of User Interface
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904098RINC
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Usability; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- User
  Interventions: Other: iOS application usability test

INTERVENTIONS:
Other: iOS application usability test — user tasks, questionnaires, semi-structured interviews

SUMMARY:
Pre-anesthesia assessment is an important part of anesthesiologists daily routine. A thorough assessment leads to an impeccable anesthesia plan. In the past, the department of anesthesiologist in NTUH (National Taiwan University Hospital) utilizes paper assessment form. As government policy leans towards digitization, the department of anesthesiologist in NTUH collaborates with the information technology office to develop an electronic pre-anesthesia assessment system called EVAN, which is an iOS based application (App). EVAN includes an anesthesia patient list, patient EMR (electronic medical record) and pre-anesthesia assessment form. EVAN was online since March, 2018.

This is an observational research to investigate the user experience and improve the user interface of EVAN.

This research subjects include anesthesiologists from NTUH. This research has three parts: user tasks, questionnaires, and a semi-structured interview. First, the research assistant will record how the user use the App to complete the tasks, which includes video recording and App monitoring. After the tasks is completed, the subject will write a questionnaire. Then the principal investigator will give an interview for feedbacks from the users.

ELIGIBILITY:
Inclusion Criteria:

* anesthesiologists in NTUH

Exclusion Criteria:

* none

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enroll the anesthesiologists and anesthesiology residents in NTUH
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
task complete time | the duration the user needs to complete the tasks, usually within 10 minutes
  the time duration the user needs to complete the user tasks

SECONDARY OUTCOMES:
questionnaire grading | after the user questionnaire completion, usually within 1 minutes
  user questionnaire grading

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No